CLINICAL TRIAL: NCT06938061
Title: Integrating 3D Imaging Technology for Precise Burn Wound Assessment
Brief Title: Utilizing 3D Imaging for Burn Wound Assessment
Status: Recruiting | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: A24-362
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Burn; 2nd Degree Burn of the Skin; 3rd Degree Burn of the Skin; 1st Degree Burn of the Skin
Keywords: 3D Imaging; AI
MeSH Terms: conditions — Burns | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 1st Degree Burn: Patients presenting to Regions Hospital Burn Clinic with a 1st degree burn
  Interventions: Device: 3D Imaging
- 2nd Degree Burn: Patients presenting to Regions Hospital Burn Clinic with a 2nd degree burn
  Interventions: Device: 3D Imaging
- 3rd Degree Burn: Patients presenting to Regions Hospital Burn Clinic with a 3rd degree burn
  Interventions: Device: 3D Imaging

INTERVENTIONS:
Device: 3D Imaging — The Derma Monitor device is a handheld, battery powered camera incorporating polarized LED illumination, a high-resolution CMOS color image sensor and a 3D depth sensor, allowing for the imaging and mapping of a patient's skin.
  Other Names: DermaMonitor Camera

SUMMARY:
The goal of this prospective cohort study is to determine if the DermaMonitor camera can accurately determine burn size in patients with 1st, 2nd, or 3rd degree burns, with exploratory aim of testing a new Artificial Intelligence (AI) program for determining burn depth. The main aims are:

1. The primary aim of this study is to assess an objective process for the classification of burn size using the DermaMonitor wound camera.
2. An exploratory aim of this study is to begin to train an Artificial Intelligence (AI) program to classify burn depth (1st, 2nd, 3rd degree) using the 3D images from this novel wound camera.

Researchers will compare DermaMonitor size classification and AI depth classification to clinician determinations. Participants will have images taken of their burn. Participation ends when the images are taken.

ELIGIBILITY:
Inclusion Criteria:

* Adults sustaining burns
* Outpatients
* No prior surgery on the wounds
* No known infection of the wounds

Exclusion Criteria:

* Burns to the face or sensitive areas (genitals)
* Burns located on or near identifying landmarks such as tattoos or birthmarks
* Non-English speaking patients
* Patients unable to sign their name
* Burn occurred greater than 7 days prior to clinic visit
* Age greater than 90 (Patient age is sent externally to IKO, to ensure no PHI is sent, patients with an age >90 will not be enrolled)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting outpatient to the Regions Hospital burn clinic after a burn
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concordance between TBSA based on Clinician measurements and TBSA based on DermaMonitor Camera measurements | Through study completion, an average of one year
  Measurements of the burn will be taken by clinicians in the burn clinic and translated into total burn surface area (TBSA) using body mass index and height. This will be compared to TBSA computed from measurements taken virtually using the DermaMonitor camera and the same body mass index and height values.

SECONDARY OUTCOMES:
Concordance between clinician burn depth determination (1st, 2nd, 3rd degree burn) and AI determination of burn depth based on DermaMonitor images | Through study completion, an average of one year
  Clinicians will subjectively determine burn depth (1st, 2nd, or 3rd degree) based on physical exam and clinical factors. This will be compared to burn depth assessment (1st, 2nd, or 3rd degree) made by an Artificial Intelligence program using the 3D images from the DermaMonitor camera.

CONTACTS AND LOCATIONS:
Locations (1):
- Regions Hospital Burn Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Consent form does not explicitly approve sharing of data with external sources.

REFERENCES:
- [Background] Irwin LR, Reid CA, McLean NR. Burns in children: do casualty officers get it right? Injury. 1993 Mar;24(3):187-8. doi: 10.1016/0020-1383(93)90291-d. PMID 8509192
- [Background] Ho HL, Halim AS, Sulaiman WAW, Fatimah MJ. Estimation of Total Body Surface Area Burned: A Comparison Between Burn Unit and Referring Facilities. Ann Burns Fire Disasters. 2023 Mar 31;36(1):19-28. eCollection 2023 Mar. PMID 38680901